CLINICAL TRIAL: NCT04203212
Title: Bone Mineral Density Alterations and Correlations With Bone and Muscle Metabolism Parameters During Menstrual Cessation Due to GnRH Therapy and After Menstrual Restoration
Brief Title: BMD Alterations and Bone and Muscle Parameters During Menstrual Cessation With GnRH
Status: Completed | Type: Observational
Sponsor: 424 General Military Hospital (Other)
Collaborators: 251 Hellenic Air Force & VA General Hospital (Other); Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Athanasios D. Anastasilakis, Consultant of endocrinology, 424 General Military Hospital
Other Study IDs: Menomyobone
Record Dates: First submitted 2019-12-15; First posted 2019-12-18 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Endometriosis; Bone Density; Muscle; Bone Metabolism
Keywords: endometriosis; bone mineral density; myokines; sclerotin; periostin
MeSH Terms: conditions — Endometriosis | interventions — Goserelin; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometriosis Group: 20 premenopausal women with surgically verified endometriosis who will receive goserelin 1 injection per month for 6 months. Subsequently goserelin will be discontinued and patients will be monitored for another 6 months after menstrual restoration.
  Interventions: Drug: Goserelin Acetate
- Control Group: 20 age- and BMI-matched premenopausal, health women who will receive no treatment and be monitored for 6 months.

INTERVENTIONS:
Drug: Goserelin Acetate — Goserelin the a GnRH analog that will be administered to achieve menstrual cessation for 6 months
  Other Names: GnRH analog
  Groups: Endometriosis Group

SUMMARY:
The investigators aim to investigate the effect of menstrual cessation in women with endometriosis treated with GnRH analogs for 6 months on bone mineral density and bone and muscle metabolism parameters and subsequently the effects of menstrual restoration after GnRH analogs discontinuation on the above measured parameters

DETAILED DESCRIPTION:
Prospective, open-label, controlled 12month observational study

Premenopausal women with surgically verified endometriosis will receive goserelin 1 injection per month for 6 months. Subsequently goserelin will be discontinued and patients will be monitored for another 6 months after menstrual restoration. Age- and BMI-matched premenopausal, health women will serve as controls. Controls will receive no treatment.

ELIGIBILITY:
Inclusion Criteria:

Premenopausal women with surgically verified endometriosis

Exclusion Criteria:

1. Secondary osteoporosis
2. diseases or conditions that could affect bone and/or muscle metabolism
3. any medications that could affect bone and/or muscle metabolism

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Premenopausal women
Study Population: Premenopausal women with surgically verified endometriosis will receive goserelin 1 injection per month for 6 months. Subsequently goserelin will be discontinued and patients will be monitored for another 6 months after menstrual restoration. Age- and BMI-matched premenopausal, health women will serve as controls
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
lumbar spine BMD | between baseline and 6 months after goserelin initiation
  Bone mineral density changes at the lumbar spine measured by dual-energy absorptiometry
lumbar spine BMD | between baseline and 6 months after goserelin discontinuation
  Bone mineral density changes at the lumbar spine measured by dual-energy absorptiometry

SECONDARY OUTCOMES:
femoral neck BMD | between baseline and 6 months after goserelin initiation
  Bone mineral density changes at the femoral neck measured by dual-energy absorptiometry
femoral neck BMD | between baseline and 6 months after goserelin discontinuation
  Bone mineral density changes at the femoral neck measured by dual-energy absorptiometry
sclerostin | 0,6,12 months
  bone metabolism parameter measured in sera
periostin | 0,3,6,12 months
  bone metabolism parameter measured in sera
irisin | 0,3,6,12 months
  myokine measured in sera
follistatin | 0,3,6,12 months
  myokine measured in sera
activin-A | 0,3,6,12 months
  myokine measured in sera
noggin | 0,3,6,12 months
  BMP inhibitor measured in sera
miRs | 0,6,12 months
  bone related microRNAs measured in sera

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Anastasilakis, PhD, Principal Investigator — 424 General Military Hospital
Locations (1):
- 424 General Military Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided
After study results being accepted for publication they will be available for everyone that might ask for them

REFERENCES:
- [Background] Paoletti AM, Serra GG, Cagnacci A, Vacca AM, Guerriero S, Solla E, Melis GB. Spontaneous reversibility of bone loss induced by gonadotropin-releasing hormone analog treatment. Fertil Steril. 1996 Apr;65(4):707-10. PMID 8654625
- [Background] Waibel-Treber S, Minne HW, Scharla SH, Bremen T, Ziegler R, Leyendecker G. Reversible bone loss in women treated with GnRH-agonists for endometriosis and uterine leiomyoma. Hum Reprod. 1989 May;4(4):384-8. doi: 10.1093/oxfordjournals.humrep.a136912. PMID 2526152
- [Background] Taga M, Minaguchi H. Reduction of bone mineral density by gonadotropin-releasing hormone agonist, nafarelin, is not completely reversible at 6 months after the cessation of administration. Acta Obstet Gynecol Scand. 1996 Feb;75(2):162-5. doi: 10.3109/00016349609033310. PMID 8604604